CLINICAL TRIAL: NCT00207285
Title: Sleep Disorders Management, Health and Safety in Police
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Charles Andrew Czeisler, MD, PhD, Charles A Czeisler, Ph.D., M.D.,, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 1R01OH008496 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Sleep Disorders; Sleep Apnea, Obstructive; Restless Legs Syndrome; Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders
Keywords: Police; Sleep; Fatigue; Work Hours; Sleep disorder; Performance
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea, Obstructive; Restless Legs Syndrome; Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Mass Screening

ARMS (3):
- In Person Training (Other): These firefighters received the sleep education and sleep disorders screening in person by one of our research staff.
  Interventions: Behavioral: Sleep Hygiene Education; Procedure: Screening and Treatment of Sleep Disorders
- Train the Trainer (Other): These firefighters received the education and sleep disorder screening in person with someone taught by our research staff.
  Interventions: Behavioral: Sleep Hygiene Education; Procedure: Screening and Treatment of Sleep Disorders
- Online Group (Other): These firefighters took the sleep disorder screening and education online.
  Interventions: Behavioral: Sleep Hygiene Education; Procedure: Screening and Treatment of Sleep Disorders

INTERVENTIONS:
Behavioral: Sleep Hygiene Education — Baseline general meetings with officers in intervention districts, in which we will provide an introductory program on optimal caffeine use (caffeine re-education) and sleep hygiene, as these are cost-effective measures that may effectively address difficulties adjusting to night work, and low-grade sleep disorders such as mild shift work sleep disorder across the cohort as a whole.
Procedure: Screening and Treatment of Sleep Disorders — All individuals who screen positive in the questionnaires on the baseline survey will be referred to one of the physicians at Sleep HealthCenters® or other sleep clinics in Massachusetts. Individuals will be paid $40 for attending an initial consultation visit with a sleep clinician and $400 if they are then asked to undergo an overnight sleep study and they complete the sleep study. Individuals will also be asked to wear an ApneaLink device for 2 nights at home and for 1 night during the overnight visit at Sleep HealthCenters®. Subjects may be asked to wear the ApneaLink device for more than 2 nights if there are not 4 hours of usable data each night. If the data is inadequate, subjects will be asked to wear the device until 4 hours of usable data on 2 nights is achieved. The ApneaLink device is an FDA approved sleep-screening tool that is used to identify individuals that are at risk for Obstructive Sleep Apnea Syndrome.

SUMMARY:
The purpose of the study is to test the effect of a sleep disorders detection and treatment program for police officers on their safety, quality of life, and job performance. The program is called Operation Healthy Sleep. We will develop and test a sleep health detection and treatment program that we aim to apply nationwide to reduce police officer fatigue and stress; enhance the ability of officers and their families to cope with police work; improve the health, safety and performance of law enforcement officers; and thereby improve public safety. Part of this program will include a questionnaire asking about about work hours and health related issues. We will then look at how these survey data relate with data on police officer safety and job performance that we are collecting through police department's databases.

Sleep disorders are common and treatable, but often remain undiagnosed and untreated. Police officers work some of the most demanding schedules known, which increases their risk of sleep disorders. The public expects officers to perform flawlessly, but unrecognized sleep disorders lead to severe disruption of sleep, which significantly reduces an individual's ability to think clearly and perform well. In addition, sleep loss and sleep disruption affect personal health, increasing the risk of gastrointestinal and cardiovascular. We also know that sleep loss increases the risk of injury due to motor vehicle crashes.

The goals of Operation Healthy Sleep are to improve officers' health, safety, and performance by reducing the impact of fatigue.

The study will take place over two years. In the first year, half of the police officers will take part in Operation Healthy Sleep, and in the second year, the second half will participate. We will carefully select the year 1 and year 2 groups so that the data collected across the two years can be validly compared.

DETAILED DESCRIPTION:
Information Session and Surveys We will visit police stations and present an information session about Operation Healthy Sleep. The session will take place during work time. During this session, we will also provide a short education session aimed to help officers to improve their sleep habits and alertness. During the session, we will invite officers to take part in Operation Healthy Sleep.

If the officer agrees to take part, he/she will be asked to provide informed consent, and then complete a survey. The survey is comprehensive and includes questions regarding work schedules, past medical history, health habits, accidents, quality of life, and mood. The survey will also include a screening test to see if they might have a sleeping disorder. The total time commitment involved in attending the information/education session and completing the survey will be about 1 to 2 hours.

Officers will be asked to provide email address and other contact information. Officers will then receive information on how to link to our monthly web-based nationwide survey. The brief monthly surveys include questions regarding work schedules, accidents and injuries, health, quality of life, and mood. The survey should take about 10-15 minutes to complete each month.

Finally, a version of the survey will be completed at the end of each year until the study is completed (i.e. at most, two years). These yearly surveys will be completed during regular work time.

During the study, we will be tracking work hours, accidents, and job performance of all officers using the police department's computerized and paper records. Data collected through this system may be compared with other data we collect from officers directly. Protection of officers' confidentiality will be our highest priority.

Assessment and Treatment of Sleep Disorders After the initial information/education session is completed, we will review responses to the survey to check whether officers are at risk of having a sleep disorder. If officers are found to be at risk, we will contact them and recommend that they undergo assessment and, if necessary, treatment by a physician or sleep specialist. We will provide the officer with referrals to local sleep disorders testing and treatment centers and physicians. Officers are free to choose another sleep disorders specialist or another physician if they prefer.

ELIGIBILITY:
Inclusion Criteria:

* Active sworn police officers

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2005-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Motor vehicle accidents as a function of miles traveled | 05/2005 - 07/2009
Number of on-the-job injuries | 05/2005 - 07/2009
Number of citations issued | 05/2005 - 07/2009
Number of arrests made | 05/2005 - 07/2009
Number of warnings issued | 05/2005 - 07/2009
Number of officer-initiated vehicle assists | 05/2005 - 07/2009
Number of sick leave days | 05/2005 - 07/2009
Sleep duration | 05/2005 - 07/2009
Sleep quality | 05/2005 - 07/2009
Alertness | 05/2005 - 07/2009
Performance | 05/2005 - 07/2009

SECONDARY OUTCOMES:
Job satisfaction | 05/2005 - 07/2009
Burnout | 05/2005 - 07/2009
Works hours | 05/2005 - 07/2009

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Czeisler, Ph.D., M.D., Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States